CLINICAL TRIAL: NCT00004398
Title: Phase I Study of Heme Arginate With or Without Tin Mesoporphyrin in Patients With Acute Attacks of Porphyria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Texas (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 199/13191; UTMB-97-118; UTMB-FDR001459
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-06

CONDITIONS: Porphyria
Keywords: inborn errors of metabolism; porphyria; rare disease
MeSH Terms: conditions — Porphyrias; Metabolism, Inborn Errors; Rare Diseases | interventions — heme arginate; tin mesoporphyrin

INTERVENTIONS:
Drug: heme arginate
Drug: tin mesoporphyrin

SUMMARY:
OBJECTIVES: I. Evaluate the efficacy of tin mesoporphyrin in patients with acute porphyria attacks who are also treated with a standard course of heme arginate.

II. Evaluate the safety and tolerability of tin mesoporphyrin when administered to these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is an randomized, unblinded, multicenter study. Patients are randomized to receive heme arginate alone or both heme arginate and tin mesoporphyrin.

Patients receive a single intravenous dose of tin mesoporphyrin immediately before the first dose of heme arginate. Heme arginate is administered daily for 4 days.

Patients are followed at 3 and 6 days after treatment.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Documented acute intermittent porphyria, variegate porphyria, or hereditary coproporphyria

No chronic or subacute symptoms (present for longer than 2 weeks)

--Prior/Concurrent Therapy--

At least 3 weeks since prior treatment with heme arginate or tin mesoporphyrin

--Patient Characteristics--

Renal: Urinary porphobilinogen at least 40 mg/24 hr

Other:

* Not pregnant
* Fertile female patients must use effective contraception during and 6 months before study
* No evidence that symptoms are due to another acute illness
* No acute hemorrhagic disorder such as: Gastrointestinal bleeding Intracerebral hemorrhage
* No known sensitivity to heme preparation or tin mesoporphyrin
* No other medical condition that might increase risk to patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 1998-01; Study Completion 2000-05

CONTACTS AND LOCATIONS:
Overall Officials: Karl Elmo Anderson, Study Chair — University of Texas